CLINICAL TRIAL: NCT06504225
Title: Long-term Evaluation of the Value of Using an MTor Inhibitor (everolimus) for the Minimisation of Anticalceurins in Old-for-old Kidney Transplantation
Brief Title: EVEROLD LONG TERM FOLLOW-UP
Acronym: EVEROLD FUP
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC23.0069 - Everold FUP
Record Dates: First submitted 2024-07-10; First posted 2024-07-16 (Actual); Last update posted 2025-02-06 (Actual); Status verified 2024-09

CONDITIONS: Transplant; Complication, Failure

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (3):
- Active Comparator: Control: Drug: Anti R-IL2 + Cyclosporine
  * Anti R-IL2 induction (Simulect ®, 20 mg D0 and D4)
  * Mycophenolate Mofetil (Cellcept ®) 3 grams per day beginning at D0
  * Cyclosporine A (Neoral ®) started from 6 to 8 mg/kg adjusted to C2
  * Corticosteroids 250 mg IV before and after surgery, then 1 mg/kg one week and 20mg/j the week after, then tapered until 10 mg/j at M1, 5 mg at M3 and stop between M4 and M6
- Experimental: CNI-free: Drug: Thymoglobulin + Everolimus
  * Thymoglobulin ® induction started at 1.5mg/kg/j then adjusted to CD2 or total lymphocytes count, for 5 days
  * Mycophenolate Mofetil (Cellcept ®) 3 grams per day beginning at D0
  * Everolimus (Certican ®): 4 to 6 mg/day started at D5, adjusted to achieve a residual level between 6 et 10 ng/ml
  * Corticosteroids 250 mg IV before and after surgery, then 1 mg/kg one week and 20mg/j the week after, then tapered until 10 mg/j at M1, 5 mg at M3 and stop between M4 and M6
- Experimental: Switch: Drug: Anti R-IL2 + Cyclosporine then Everolimus
  * Anti R-IL2 induction (Simulect ®, 20 mg D0 and D4)
  * Mycophenolate Mofetil (Cellcept ®) 3 g/d beginning at D0
  * Cyclosporine A (Neoral ®) beginning at 6 to 8 mg/kg adjusted to C2, then switch to everolimus (Certican ®) between at W6, started at 3 mg/d, then adjusted to achieve a residual level between 6 et 10 ng/ml
  * Corticosteroids 250 mg IV before and after surgery, then 1 mg/kg one week and 20mg/j the week after, then tapered until 10 mg/j at M1, 5 mg at M3 and stop between M4 and M6

SUMMARY:
Long Term Follow up of EVEROLD study

ELIGIBILITY:
Inclusion Criteria:

* Informed patients participating to the EVEROLD study
* Patient having completed the EVEROLD M12 follow-up visit
* Patient agreeing to participate in the observational study

Exclusion Criteria:

* Opposition to the use his medical data
* Patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 260 patients previously included in the EVEROLD study
Sampling Method: Non-Probability Sample
Enrollment: 260 (Estimated)
Dates: Start 2024-08-23 (Actual); Primary Completion 2025-08-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Patient survival | up to 12 years
  Patient survival at last follow-up
Graft survival | up to 12 years
  Graft survival at last follow-up

SECONDARY OUTCOMES:
Rejection rate | up to 12 years
  Biopsy proven rejection
Infection rate | up to 12 years
  All infections requiring hospitalization
Major cardiovascular events | up to 12 years
Cancer rate | up to 12 years
  Skin cancer, solid organ tumor and hematological cancer
Hospitalization | up to 12 years
  Number of hospitalization, hospital stay, reason for hospitalization
eGFR | up to 12 years
  estimated GFR (MDRD and CKD-EPI)

CONTACTS AND LOCATIONS:
Overall Officials: Yannick LE MEUR, Principal Investigator — CHU Brest
Locations (14):
- France (14):
  - Chu Amiens, Amiens
  - CHU Bordeaux, Bordeaux
  - Chu Brest, Brest
  - CHU Lille, Lille
  - CHU Limoges, Limoges
  - CHU Nice Pasteur 2, Nice
  - CHU Nice, Nice
  - Hôpital Necker, Paris
  - Chu Poitiers, Poitiers
  - CHU Rennes, Rennes
  - CHU Rouen, Rouen
  - CHU Strasbourg, Strasbourg
  - CHU Toulouse Rangueil, Toulouse
  - CHU Tours, Tours

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement